CLINICAL TRIAL: NCT03079167
Title: Preventing Adverse Outcomes of Neonatal Hypoxic Ischaemic Encephalopathy With Erythropoietin: A Phase III Randomised Placebo Controlled Multicentre Clinical Trial
Brief Title: PAEAN - Erythropoietin for Hypoxic Ischaemic Encephalopathy in Newborns
Acronym: PAEAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTC0119; 12614000669695 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2017-02-20; First posted 2017-03-14 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Epoetin Alfa; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin (Experimental): Erythropoietin (epoetin alfa) 1000 IU/kg birth weight (capped at 4000IU daily) IV infusion, on Days 1, 2, 3, 5 and 7 of age
  Interventions: Drug: Epoetin Alfa
- Placebo (Placebo Comparator): IV normal saline (equiv. volume), on Days 1, 2, 3, 5 and 7 of age
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Epoetin Alfa
  Other Names: Epogen; Procrit
  Arms: Erythropoietin
Drug: Normal saline
  Other Names: 0.9% NaCl
  Arms: Placebo

SUMMARY:
Double-blind, placebo controlled Phase III trial of erythropoietin for hypoxic ischaemic encephalopathy in infants receiving hypothermia. The study aim is to determine whether Epo in conjunction with hypothermia in infants with moderate/severe hypoxic ischaemic encephalopathy (HIE) will improve neurodevelopmental outcomes at 2 years of age, without significant adverse effects, when compared to hypothermia alone.

DETAILED DESCRIPTION:
A lack of oxygen (hypoxia) or low blood supply (ischaemia) before or during birth can destroy cells in a newborn baby's brain. The damage caused by the lack of oxygen continues for some time afterwards. One way to try to reduce this damage is to induce hypothermia cooling the baby or just the baby's head for hours to days. Erythropoietin (Epo) given in the first week after birth shows promise as a treatment that may also help. This study is to find out whether Epo plus induced hypothermia (cooling) of near-term newborn babies who have suffered from low blood or oxygen supply to the brain at birth reduces death and disability in survivors at two years of age.

The target population is 300 newborn term or near term infants (greater than or equal to 35+0 weeks gestation) with hypoxic ischaemic encephalopathy who are receiving, or planned to receive hypothermia and who are able to be recruited in time to allow study treatment to commence before 24 hours of age.

This is a double blind, placebo controlled, parallel, 2 arm randomised, phase III multicentre trial, stratified by study site and by severity of encephalopathy at study entry.

The treatment group of 150 infants will receive human recombinant Epo, 1000 IU/kg IV on days 1, 2, 3, 5 & 7 of life. The control group will receive 0.9% sodium chloride as a placebo on days 1, 2, 3, 5 & 7 of life.

Families will be followed up every 6 months until the primary assessment of death and disability at 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants born greater than or equal to 35+0 weeks gestation and able to be randomised less than 23 hours after birth
* One or more of the following indicators of perinatal depression:

  1. Apgar less than or equal to 5 at 10 minutes after birth, OR
  2. Receiving ongoing resuscitation e.g. assisted ventilation (positive pressure ventilation or CPAP) or chest compressions at 10 minutes after birth, OR
  3. on cord blood or arterial or venous blood obtained at less than 60 minutes after birth, either pH less than 7.00 OR base deficit greater than or equal to 12.0 mmol/L
* Moderate to severe encephalopathy, defined between one and six hours after birth by one or both of the following:

  1. 3 out of 6 modified Sarnat criteria indicating moderate/severe encephalopathy, OR
  2. 2 out of 6 modified Sarnat criteria plus seizure(s) requiring anticonvulsant treatment (diagnosed either clinically or using EEG monitoring) at any time prior to randomisation
* Hypothermia treatment initiated by 6 hours ofa ge; i.e. controlled whole-body cooling planned to continue for 72 hours to a target temperature (adjusted manually or with a device) and subsequent controlled re-warming
* Study treatment planned to start within 24 hours after birth (as soon as feasible after randomisation)
* At least one parent greater than or equal to 18 years of age
* Anticipated ability to collect primary endpoint at 2 years of age
* Signed, written informed parental consent

Exclusion Criteria:

* Contraindications to investigational product
* Indication prior to randomisation for erythropoietin or any other erythropoietic stimulating agent to be given during the first two weeks of life
* Severe intrauterine growth restriction (birth weight less than 1800g)
* Suspected major chromosomal or congenital anomalies
* Head circumference less than 3rd centile below the mean for gestation and gender
* Infant for whom imminent withdrawal of care is being planned

Max Age: 23 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 313 (Actual)
Dates: Start 2016-05-14 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Composite measure of death or moderate/severe disability | 2 years of age
  Moderate/severe disability is defined as any cerebral palsy and a Gross Motor Function Classification Scale (GMFCS) score greater than or equal to 1), or Bayley Scale of Infant Development III (BSDIII) less than or equal to 80

SECONDARY OUTCOMES:
Death | Any time from Day 1 of treatment to 2 years of age
  Death from any cause
Cerebral palsy (CP), assessed by paediatric assessment | 2 years of age
  Any incidence of CP (any of quadriplegia, triplegia, hemiplegia, diplegia or monoplegia)
Moderate/severe motor deficit | 2 years of age
  Composite of any incidence of CP (any of quadriparesis, CP, hemiparesis or diparesis) AND any level of functional impairment using the GMFCS greater than or equal to 1.0
Moderate/severe cognitive deficit | 2 years of age
  Defined as a BSDIII cognitive score less than or equal to 80
Need for supplemental respiratory support (includes tracheostomy, ventilator, high flow nasal cannula, CPAP or oxygen dependency) | 2 years of age
  Supplemental respiratory support includes tracheostomy, ventilator, high flow nasal cannula, CPAP or oxygen dependency
Need for nutritional support (includes gastrostomy or nasogastric feeds) | 2 years of age
  Nutritional support includes gastrostomy or nasogastric feeds
Major cortical visual impairment by paediatric examination | 2 years of age
  Impairment as assessed by paediatric assessment
Hearing impairment status by paediatric examination - requirement for hearing aids | 2 years of age
  Defined as the requirement for hearing aids (either diagnosis of: Hears well or with only a little difficulty WITH a hearing aid OR Has severe hearing difficulty even with a hearing aid or hearing is not helped with an aid)
Epilepsy (history of 2 or more afebrile unprovoked seizures since discharge from neonatal unit where PAEAN study treatment was provided, or use of anticonvulsants at 2 years of age). | 2 years of age
  Defined by history of 2 or more afebrile unprovoked seizures since discharge from neonatal unit where PAEAN study treatment was provided, or use of anticonvulsants at 2 years of age
Cost of healthcare and service utilisation | 2 years of age
  Defined as a composite of parent completed questionnaire data and Medicare service use
Frequency of selected adverse events (AEs) of interest, including deaths | Up to 30 days post study treatment
  Frequency of selected adverse events (AEs) of interest up to 30 days after the last study dose

OTHER OUTCOMES:
Distribution of overall disability | 2 years of age
  Distribution of overall severity across 4 domains: 1) normal, 2) mild motor or cognitive deficit, 3) moderate/severe motor or cognitive deficit, and 4) death

CONTACTS AND LOCATIONS:
Overall Officials: Helen Liley, BHB, MBChB, Study Chair — University of Sydney
Locations (24):
- Australia (18):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal Hospital for Women, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Women's & Brisbane Hospital, Herston, Queensland
  - Mater Mothers' Hospital, South Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - Mercy Hospital for Women, Heidelberg, Victoria
  - The Royal Children's Hospital, Parkville, Victoria
  - The Royal Women's Hospital, Parkville, Victoria
  - King Edward Memorial Hospital, Subiaco, Western Australia
  - Princess Margaret Hospital, Subiaco, Western Australia
- New Zealand (5):
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No